CLINICAL TRIAL: NCT04071210
Title: Impact of Oral Probiotics on Oral Homeostasis - a Randomized Double Blind Study
Brief Title: Impact of Oral Probiotics on Oral Homeostasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Daniel Belstrøm, DDS, PhD, Associate professor, Principal Investiator, dr. odont., PhD, DDS, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UCPH_OI_003
Record Dates: First submitted 2019-08-19; First posted 2019-08-28 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Randomized double blind clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: PI are the only one aware of participant status.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Probiotic tablets (containing a mix of Lactobacillus rhamnosus PB01, DSM 14869 and Lactobacillus curvatus EB10, DSM 32307, 1*10(9) CFU) 2 times/day for 12 weeks
  Interventions: Dietary Supplement: Probiotic tablet
- Placebo Comparator (Placebo Comparator): Placebo tablets 2 times/day for 12 weeks
  Interventions: Dietary Supplement: Placebo tablet

INTERVENTIONS:
Dietary Supplement: Probiotic tablet — Probiotic tablet twice a day for 12 weeks
  Arms: Experimental
Dietary Supplement: Placebo tablet — Placebo tablet twice a day for 12 weeks
  Arms: Placebo Comparator

SUMMARY:
Aim:

To evaluate the effect of three months use of tablets containing probiotics on the composition of the supragingival plaque microbiota and salivary levels of inflammation-related proteins in oral healthy individuals.

Hypothesis:

Three months use of tablets containing probiotics will induce quantifiable changes to the composition of the supragingival plaque microbiota and salivary levels of inflammation-related proteins in oral healthy individuals.

Perspectives:

Data from the present study will be able to reveal the impact of regular use of probiotics on oral homeostasis in oral healthy individuals. Specifically, simultaneous registration of clinical, microbial and inflammatory characteristics will provide comprehensive information on the potential beneficial effect of regular use of oral probiotics on maintenance of oral homeostasis. Thus, data from the present study will provide a scientific platform, which dentist and dental hygienist can utilize when deciding if oral healthy individuals may benefit from using oral probiotics as a supplement to regular oral hygiene.

DETAILED DESCRIPTION:
Oral health is built upon a symbiotic relationship between the resident oral microbiota and the immune system of the host. Therefore, structural or functional changes to either the microbiota or the immune system may result in dysbiosis, which in turn can lead to oral diseases such as gingivitis, periodontitis and dental caries.

The composition of the resident oral microbiota in oral health is shaped by ecological properties found at various sites of the oral cavity, which is why major site-specific variations are observed. Interestingly, the composition of the oral microbiota is individualized and relatively time stable as long as oral homeostasis is maintained. However, structure and function of the oral microbiota can be altered by internal and external perturbations. For example, it has previously demonstrated that oral hygiene discontinuation induces structural changes to the supragingival plaque microbiota, whereas non-surgical periodontal treatment has deep impact on the composition of the subgingival plaque microbiota. Interestingly, a recent study demonstrated that the composition of the resident oral microbiota may also be influenced by external perturbations. Specifically, daily use of ZendiumTM toothpaste for 12 weeks was reported to induce significant changes to the supragingival plaque microbiota in oral healthy individuals with an increase in health-associated bacterial species.

Probiotics is the term used when a harmless effector strain is implanted in the host's microbiota to maintain or restore a natural microbiome by interference and/or inhibition of other microorganisms, and especially pathogens. In a recent study, it was demonstrated an effect of using tablets containing a mix of Lactobacillus rhamnosus PB01, DSM 14869 and Lactobacillus curvatus EB10, DSM 32307 on gingival inflammation. Specifically, daily use of this probiotic candidate for four weeks resulted in significant reduction in clinical parameters such as bleeding on probing (BOP) and amount of gingival crevicular fluid (GCF).

However, at present it is not known if daily use of a probiotic tablet containing a mix of L. rhamnosus PB01, DSM 14869 and L. curvatus EB10, DSM 32307 is able to induce shifts to the composition of the oral microbiota, or cause a decrease in salivary levels of inflammation-related proteins such as neutrophil gelatinase-associated lipocalin (NGAL) and transferrin, which is the purpose of the present study.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 yrs.

Exclusion Criteria:

* gingivitis
* periodontitis
* dental caries
* systemic disease
* current medication
* antibiotic treatment within the latest 3 months.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Change in bacterial diversity of supragingival plaque microbiota from baseline to week 12 | Baseline alpha-diversity vs. alpha-diversity at week 12
  Alpha-diversity measured by shannon index

SECONDARY OUTCOMES:
Change in salivary levels of neutrophil gelatinase-associated lipocalin (NGAL) from baseline to week 12 | Baseline levels vs. leves at week 12.
  Mean levels of NGAL (mg/mL) measured by ELISA
Change in Salivary levels of transferrin from baseline to week 12 | Baseline levels vs. leves at week 12.
  Mean levels of transferrin (mg/mL) measured by ELISA

OTHER OUTCOMES:
Change in plaque index (PI) from baseline to week 12 | Baseline recordings vs. recordings at week 12.
  Mean levels of PI (% of sites with positive recordings)
Change in gingival inflammation index (GI) from baseline to week 12 | Baseline recordings vs. recordings at week 12.
  Mean levels of GI (% of sites with positive recordings)
Change in bleeding index (BI) from baseline to week 12 | Baseline recordings vs. recordings at week 12.
  Mean levels of BI (% of sites with positive recordings)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Copenhagen, Dept. of Odontology, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No